CLINICAL TRIAL: NCT00876980
Title: The Effect of Nasal Continuous Positive Airway Pressure Treatment on Glycemic Control and Vascular Function in Patients With Obstructive Sleep Apnea and Type II Diabetes Mellitus.
Brief Title: Obstructive Sleep Apnea and Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lam Jamie Chung Mei, Honorary clinical assistant professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKCTR-676
Record Dates: First submitted 2009-03-23; First posted 2009-04-07 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Obstructive Sleep Apnea; Diabetes Mellitus
Keywords: Obstructive sleep apnea; Type II diabetes mellitus; Randomized controlled trial
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): nasal Continuous Positive Airway Pressure treatment for 3 months
  Interventions: Device: nasal Continuous Positive Airway Pressure
- 2 (No Intervention): controls have no treatment, being observed for 3 months

INTERVENTIONS:
Device: nasal Continuous Positive Airway Pressure — A standard treatment for OSA. A portable machine delivers positive pressure through a mask to the upper airway during sleep at night.
  Other Names: nCPAP
  Arms: 1

SUMMARY:
The investigators hypothesize that obstructive sleep apnea (OSA) contributes to impaired glucose homeostasis and associated vasculopathy, and nCPAP treatment of OSA should improve glycemic control and vascular function in OSA patients with type II diabetes mellitus. This study aims to investigate the therapeutic effects of nCPAP on glycemic control and vascular function in patients with OSA and type II diabetes mellitus.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) has been reported to be common (17%) in patients with diabetes mellitus (DM). Both OSA and DM are highly associated with cardiovascular morbidity and mortality. There is growing evidence that OSA may trigger or worsen pre-existing adverse metabolic profile indicative of cardiovascular risk. Treatment of OSA with nasal Continuous Positive Airway Pressure (nCPAP) has been shown to reduce blood pressure and hence to reduce the risk of atherogenesis. In patients with DM, the therapeutic effect of nCPAP is still not known, it would be important to delineate any independent effect of OSA on DM and the therapeutic effect of nCPAP on glycemic control to reduce the long term risk of macrovascular and microvascular complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type II DM on a stable medication regimen (on diet / oral hypoglycaemic agents / insulin injections)
2. Age 25 - 70 years
3. HbA1C > 7%
4. AHI >= 15
5. Able to give written informed consent

Exclusion Criteria:

1. Patients with severe co-existing illness or poor functional performance
2. Patients with peripheral vascular diseases, vasculitis / Raynaud's syndrome or thrombocytopenia
3. Sleep disorders other than OSA
4. Patients who refuse nCPAP treatment for OSA
5. Excessive sleepiness causing potential harm (e.g. driver)
6. HbA1C >=7%
7. Habitual drinker (defined as more than 3 times a week)
8. Pregnant or lactating women

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
HbA1C | 3 months

SECONDARY OUTCOMES:
Fasting glucose & fructosamine microalbuminuria blood pressure lipids endothelial function | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Ip, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, University Department of Medicine, Pokfulam, Hong Kong, Hong Kong

REFERENCES:
- [Result] West SD, Nicoll DJ, Wallace TM, Matthews DR, Stradling JR. Effect of CPAP on insulin resistance and HbA1c in men with obstructive sleep apnoea and type 2 diabetes. Thorax. 2007 Nov;62(11):969-74. doi: 10.1136/thx.2006.074351. Epub 2007 Jun 8. PMID 17557769